CLINICAL TRIAL: NCT00606047
Title: Prevalence of Femoroacetabular Impingement in Asymptomatic Patients
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-813
Record Dates: First submitted 2008-01-21; First posted 2008-02-01 (Estimated); Results first posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Femoroacetabular Hip Impingement Syndrome
Keywords: femoroacetabular impingement
MeSH Terms: conditions — Femoracetabular Impingement | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Asymptomatic patients: Asymptomatic, healthy patients (without hip pain or prior hip disease) will be recruited. Patients will undergo a magnetic resonance imaging (MRI) of the hip joints to evaluate for the prevalence of femoroacetabular impingement (FAI).
  Interventions: Radiation: Magnetic resonance imaging (MRI)

INTERVENTIONS:
Radiation: Magnetic resonance imaging (MRI) — Participation in this study will involve patients coming to the hospital after regular work hours for an MRI of the hip joints.

SUMMARY:
Femoroacetabular hip impingement syndrome is a newly recognized cause of early arthritis of the hip. In this condition a variation in the shape of the upper thigh bone causes it to repeatedly come in contact with the hip socket leading to cartilage damage and arthritis. The purpose of this study is to investigate whether patients without hip pain have variations at the hip joint such as those seen in hip impingement syndrome.

DETAILED DESCRIPTION:
Participants in this study will be asked to come to the hospital after regular work hours for an MRI of the hip joints. Prior to the MRI, a physician will perform a range of motion check of the participants hips. The MRI will take approximately 20 minutes during which the participant will have to lie still in a closed space. Participants will receive a letter which can be forwarded to their family doctor if the MRI has any abnormal findings including signs of hip impingement.

ELIGIBILITY:
Inclusion Criteria:

* No hip problems
* No containdications to MRI

Exclusion Criteria:

- Patient does not meet above criteria

Max Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2007-08-01 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Beaulé, MD, FRCSC, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Result] Khanna V, Caragianis A, Diprimio G, Rakhra K, Beaule PE. Incidence of hip pain in a prospective cohort of asymptomatic volunteers: is the cam deformity a risk factor for hip pain? Am J Sports Med. 2014 Apr;42(4):793-7. doi: 10.1177/0363546513518417. Epub 2014 Jan 30. PMID 24481825
- [Result] Hack K, Di Primio G, Rakhra K, Beaule PE. Prevalence of cam-type femoroacetabular impingement morphology in asymptomatic volunteers. J Bone Joint Surg Am. 2010 Oct 20;92(14):2436-44. doi: 10.2106/JBJS.J.01280. PMID 20962194

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Asymptomatic Patients
Started | 200
Completed | 200
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Asymptomatic Patients
Number analyzed (Participants) | 200
Age, Continuous [Mean (Full Range); unit: years] | 29.4 [21.4 to 50.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111
  Male | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 197
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 200
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.49 (3.18)
Handedness [Count of Participants; unit: Participants]
  Left-handedness | 12
  Right-handedness | 188
Family History of Hip Osteoarthritis [Count of Participants; unit: Participants]
  None | 184
  Family History of Hip Osteoarthritis | 16
Personal History of Childhood Hip Problems [Count of Participants; unit: Participants]
  None | 200
  Personal History of Childhood Hip Problems | 0

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Femoroacetabular Impingement (FAI)
Description: Prevalence of femoroacetabular impingement (FAI), a newly recognized cause of early arthritis of the hip, will be investigated by means of hip MRI to evaluate for abnormal morphology of the anterior head-neck junction of the femur. Participant MRIs were reviewed by two independent radiologists. The prevalence of FAI was calculated as determined by an abnormal alpha angle (greater than 50.5 degrees).
Time Frame: Pre-operative on Day of MRI
Measure: Count of Participants; unit: Participants
Arm/Group | Asymptomatic Patients
Number analyzed (Participants) | 200
Participants
  Prevalence of Cam-Type FAI | 28
  No prevalence | 172

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Asymptomatic Patients
All-Cause Mortality (participants affected / at risk) | 0/200
Serious Adverse Events (participants affected / at risk) | 0/200
Other Adverse Events (participants affected / at risk) | 0/200

LIMITATIONS AND CAVEATS:
A limitation of our study sample is that it may not truly represent the normal population as it was based in a hospital setting. However, the hospital where this study was conducted employs over 13,000 individuals with a varied work force.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2006-12-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT00606047/Prot_SAP_000.pdf